CLINICAL TRIAL: NCT04452279
Title: Prospective Study of Ocular Surface Disease Changes After iStent or iStent Inject Trabecular Micro-Bypass Implantation With Cataract Surgery
Brief Title: Ocular Surface Disease Changes After iStent or iStent Inject Implantation With Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The OSD iStent Study
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Ocular Surface Disease; Glaucoma, Open-Angle
Keywords: ocular surface; dry eye; medication; quality of life
MeSH Terms: conditions — Glaucoma, Open-Angle; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ocular Surface Disease post-stenting (Experimental): Eyes will undergo phacoemulsification cataract surgery combined with iStent or iStent inject implantation according to standard clinical practice. From baseline through 3 months postoperatively, participants will complete subjective and objective assessments of ocular surface disease.
  Interventions: Device: iStent or iStent inject implantation with concomitant cataract surgery

INTERVENTIONS:
Device: iStent or iStent inject implantation with concomitant cataract surgery — Standard phacoemulsification cataract surgery followed by ab interno implantation of either iStent or iStent inject trabecular micro-bypass stent(s). Preoperatively and at specified visits through 3 months postoperative, patients will complete evaluations of their ocular surface disease (specifically OSDI score, hyperemia, corneal/conjunctival staining, and tear break-up time).
  Other Names: iStent or iStent inject

SUMMARY:
This prospective interventional single-arm trial evaluates measures changes in ocular surface disease parameters in eyes with mild to moderate open-angle glaucoma (OAG) on 1-4 glaucoma medications who undergo phacoemulsification and trabecular micro-bypass stent(s) implantation (iStent or iStent inject).

DETAILED DESCRIPTION:
This study enrolled eyes with mild to moderate open-angle glaucoma (OAG) on 1-4 glaucoma medications who were scheduled to undergo phacoemulsification cataract extraction and trabecular micro-bypass stent(s) implantation (iStent or iStent inject). Study participation entailed measurement of key ocular surface data through 3 months postoperative including Ocular Surface Disease Index score (OSDI), corneal/conjunctival staining (Oxford Schema), fluorescein tear break-up time (FTBUT), and conjunctival hyperemia (Efron Scale); these measures were collected alongside standard postoperative glaucoma evaluations such as number of glaucoma medications and intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate primary open-angle glaucoma
2. Currently treated with ocular hypotensive medication
3. Primary open-angle, pseudoexfoliative and pigmentary glaucoma are acceptable diagnoses
4. Subject scheduled to undergo cataract surgery in combination with one trabecular meshwork bypass stent
5. 22 years of age or older
6. Able and willing to attend scheduled follow-up exams for three months postoperatively
7. Able and willing to provide written informed consent on the IRB approved Informed Consent Form
8. Successful, uncomplicated cataract surgery
9. OSDI of 8 or more

Exclusion Criteria:

* 1. Primary angle-closure glaucoma; or secondary angle closure glaucoma, including neovascular glaucoma 2. Any pathology for which, in the investigator's judgement, the following would be either at risk or contraindicated:

  1. Cataract surgery
  2. Stent implantation
  3. Compliance to elements of the study protocol (e.g., ophthalmic examinations, follow-up visits) 3. Fellow eye actively enrolled in this trial 4. Current participation in any study, or participation within 30 calendar days of screening exam 5. Unsuccessful, complicated cataract surgery 6. OSDI of 7 or less

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Change in mean OSDI score | 3 months
  Difference between preoperative and Month 3 mean OSDI score
Change in mean conjunctival hyperemia score | 3 months
  Difference between preoperative and Month 3 mean Efron score of conjunctival hyperemia
Change in mean corneal/conjunctival staining score | 3 months
  Difference between preoperative and Month 3 mean Oxford score of corneal/conjunctival hyperemia
Change in mean fluorescein tear break-up time (FTBUT) | 3 months
  Difference between preoperative and Month 3 mean FTBUT in seconds

SECONDARY OUTCOMES:
IOP change | 3 months
  Difference between preoperative and Month 3 mean IOP in mmHg
Medication change | 3 months
  Difference between preoperative and Month 3 mean number of glaucoma medications

CONTACTS AND LOCATIONS:
Overall Officials: Justin Schweitzer, OD, FAAO, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schweitzer JA, Hauser WH, Ibach M, Baartman B, Gollamudi SR, Crothers AW, Linn JE, Berdahl JP. Prospective Interventional Cohort Study of Ocular Surface Disease Changes in Eyes After Trabecular Micro-Bypass Stent(s) Implantation (iStent or iStent inject) with Phacoemulsification. Ophthalmol Ther. 2020 Dec;9(4):941-953. doi: 10.1007/s40123-020-00290-6. Epub 2020 Aug 13. PMID 32789800